CLINICAL TRIAL: NCT00416715
Title: A Pilot Study of Vitamin D Deficiency and Myalgias, Arthralgias and/or Joint Stiffness Associated With Letrozole (Femara® )
Brief Title: Vitamin D Deficiency, Muscle Pain, Joint Pain, and Joint Stiffness in Postmenopausal Women Receiving Letrozole For Stage I-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6346; NCI-2010-00621 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Arthralgia; Musculoskeletal Complications; Pain; Recurrent Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Arthralgia; Pain; Breast Neoplasms | interventions — Letrozole; Calcium Carbonate; Calcium Citrate; Glucaric Acid; Calcium Gluconate; Calcium; Cholecalciferol; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (letrozole) (Experimental): Patients receive letrozole PO QD. Patients, who experience muscle pain, joint pain, or joint stiffness that requires an intervention and who are found to be vitamin D deficient, also receive calcium and vitamin D3 PO. Treatment continues for up to 28 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: letrozole; Dietary Supplement: calcium carbonate; Other: laboratory biomarker analysis; Dietary Supplement: calcium citrate; Dietary Supplement: calcium glucarate; Drug: calcium gluconate; Dietary Supplement: cholecalciferol; Procedure: assessment of therapy complications; Procedure: musculoskeletal complications management/prevention

INTERVENTIONS:
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Dietary Supplement: calcium carbonate — Given PO
  Other Names: CaCO3
Other: laboratory biomarker analysis — Optional correlative studies
Dietary Supplement: calcium citrate — Given PO
  Other Names: Acicontral; CALCIT; Citracal; Tricalcium Citrate
Dietary Supplement: calcium glucarate — Given PO
  Other Names: antacidin; calcium D-glucarate; calcium D-saccharate; CGT
Drug: calcium gluconate — Given PO
  Other Names: Calcium D-gluconate; CALGLUC; Calglucon
Dietary Supplement: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3
Procedure: assessment of therapy complications — Ancillary studies
Procedure: musculoskeletal complications management/prevention — Correlative studies
  Other Names: complications management/prevention, musculoskeletal; management/prevention, musculoskeletal complications

SUMMARY:
This phase II trial is studying vitamin D deficiency, muscle pain, joint pain, and joint stiffness in postmenopausal women receiving letrozole for stage I-III breast cancer. Learning about vitamin D deficiency and muscle pain, joint pain, and joint stiffness in patients receiving letrozole for breast cancer may help doctors plan treatment and may help patients live more comfortably

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of vitamin D deficiency in breast cancer patients who experience myalgias, arthralgias and/or joint stiffness following initiation of adjuvant letrozole treatment.

SECONDARY OBJECTIVES:

I. To determine if there is a correlation between letrozole serum levels and the development of myalgias, arthralgias and/or joint stiffness.

II. To assess if vitamin D supplementation may alleviate myalgias, arthralgias and/or joint stiffness associated with letrozole in those subjects with vitamin D deficiency.

OUTLINE:

Patients receive letrozole orally (PO) once daily (QD). Patients, who experience muscle pain, joint pain, or joint stiffness that requires an intervention and who are found to be vitamin D deficient, also receive calcium PO and vitamin D3 PO. Treatment continues for up to 28 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of Stage I, II or III breast carcinoma
* Patients must be prescribed letrozole for adjuvant breast cancer treatment
* Prior adjuvant tamoxifen is permitted
* Patients must be postmenopausal; for study purposes, postmenopausal is defined as: a prior documented bilateral oophorectomy, or a history of at least 12 months without spontaneous menstrual bleeding, or have a persistently postmenopausal estradiol in the past 6 months without menses, and clinically in menopause at the judgment of the treating physician, or age 60 or older with a prior hysterectomy without oophorectomy, or age less than 60 with a prior hysterectomy without oophorectomy (or in whom the status of the ovaries is unknown), with a documented FSH level demonstrating confirmatory elevation in the postmenopausal range for the lab

Exclusion Criteria:

* Diagnosis of Stage IV breast carcinoma
* Pre-existing myalgias, arthralgias and/or joint stiffness >= Grade 1, as defined using CTEP CTC identified during baseline physical exam
* Inability to understand or cooperate with study procedures
* Receipt of investigational drug within 30 days before study entry
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Unwillingness to give informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Patients with serum calcium >= 14 mg/dL
* Patients with renal dysfunction defined as glomerular filtration rate <10ml/min calculated using Cockroft-Gault equation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Letrozole): Patients receive letrozole PO QD. Patients, who experience muscle pain, joint pain, or joint stiffness and who are found to be vitamin D deficient, also receive calcium and vitamin D3 PO. Treatment continues for up to 28 weeks in the absence of disease progression or unacceptable toxicity.
  letrozole: Given PO
  calcium carbonate: Given PO
  laboratory biomarker analysis: Optional correlative studies
  calcium citrate: Given PO
  calcium glucarate: Given PO
  calcium gluconate: Given PO
  cholecalciferol: Given PO
  assessment of therapy complications: Ancillary studies
  musculoskeletal complications management/prevention: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Letrozole)
Started | 100
Completed | 85
Not Completed | 15
Not completed — Not evaluable for joint aches | 7
Not completed — Vitamin D levels not evaluable | 8

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Letrozole)
Number analyzed (Participants) | 100
Age, Continuous [Median (Full Range); unit: years] | 56 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 87
  More than one race | 3
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Early Breast Cancer Patients Prescribed Adjuvant Letrozole That Are Vitamin D Deficient and Who Experience Myalgias, Arthralgias and/or Joint Stiffness
Description: Count of early breast cancer patients prescribed adjuvant letrozole that are vitamin D deficient and who experience myalgias, arthralgias and/or joint stiffness, assessed at baseline and 1 month after vitamin D repletion.
Time Frame: Baseline and 1 month post vitamin D repletion
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: All patients that are evaluable for joint aches and vitamin D levels.
- Post Vitamin D Repletion (1 Month): Patients with vitamin D deficiency who experience myalgias, arthralgias and/or joint stiffness.
Arm/Group | Baseline | Post Vitamin D Repletion (1 Month)
Number analyzed (Participants) | 85 | 12
Participants | 12 | 1

2. Secondary Outcome: Letrozole Serum Levels Before and After Vitamin D Repletion
Description: Letrezole serum level concentration in patients that were vitamin D deficient and experienced myalgias, arthralgias and/or joint stiffness.
Time Frame: Baseline and 1 month post vitamin D repletion
Population: Only considering those patients who were baseline vitamin D deficient and experienced myalgias, arthralgias and/or joint stiffness.
Measure: Median (Inter-Quartile Range); unit: micro-grams/mL
Groups:
- Baseline: Those receiving Letrozole + vitamin D3
- Post Vitamin D Repletion (1 Month): Those receiving Letrezole + vitamin D3
Arm/Group | Baseline | Post Vitamin D Repletion (1 Month)
Number analyzed (Participants) | 12 | 12
micro-grams/mL | 85 [63 to 100] | 70 [69 to 105]

ADVERSE EVENTS:
Groups:
- Treatment (Letrezole): Patients receive letrozole PO QD. Patients, who experience muscle pain, joint pain, or joint stiffness and who are found to be vitamin D deficient, also receive calcium and vitamin D3 PO. Treatment continues for up to 28 weeks in the absence of disease progression or unacceptable toxicity.
  letrozole: Given PO
  calcium carbonate: Given PO
  laboratory biomarker analysis: Optional correlative studies
  calcium citrate: Given PO
  calcium glucarate: Given PO
  calcium gluconate: Given PO
  cholecalciferol: Given PO
  assessment of therapy complications: Ancillary studies
  musculoskeletal complications management/prevention: Correlative studies
Arm/Group | Treatment (Letrezole)
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 27/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Letrezole) (N=100)
Joint aches (General disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes